CLINICAL TRIAL: NCT01683552
Title: Aprepitant in the Management of Biological Therapies-related Severe Pruritus: a Pilot Study in 45 Cancer Patients
Brief Title: Aprepitant in the Management of Biological Therapies-related Severe Pruritus
Acronym: AprepIt
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Daniele Santini, MD, PhD, Campus Bio-Medico University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Aprepitant-Itch
Record Dates: First submitted 2012-09-05; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: ITCH
Keywords: ITCH
MeSH Terms: interventions — Aprepitant; Prednisone; fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Other): Aprepitant is administered in patients ,affected by solid tumors treated with biological therapy, who did not receive any treatment for severe pruritus
  Interventions: Drug: Aprepitant
- Aprepitant after anti-itch standard therapy (Other): Aprepitant will be administered in patient affected by severe itch resistant to standard treatment (steroids and/or antihistamines) administered for at least one week
  Interventions: Drug: Aprepitant; Drug: Prednisone; Drug: Fexofenadine

INTERVENTIONS:
Drug: Aprepitant — 125 mg on day 1; 80 mg on day 3; 80 mg on day 5
  Other Names: Emend
Drug: Prednisone — In the refractory group (VAS score ≥7), Aprepitant (125 mg on day 1; 80 mg on day 3; 80 mg on day 5) is administered after at least one week of standard systemic treatment (prednisone 25 mg/die and/or fexofenadine 180 mg/die),
  Arms: Aprepitant after anti-itch standard therapy
Drug: Fexofenadine — In the refractory group (VAS score ≥7), Aprepitant (125 mg on day 1; 80 mg on day 3; 80 mg on day 5) is administered after at least one week of standard systemic treatment (prednisone 25 mg/die and/or fexofenadine 180 mg/die)
  Arms: Aprepitant after anti-itch standard therapy

SUMMARY:
Itch is a common side effect of anti-epidermal growth factor receptor antibodies and tyrosine kinase inhibitors. Investigators designed a pilot single-center phase II study evaluating the effects of Aprepitant, a neurokinin receptor inhibitor, in managing biological therapy-induced pruritus.

DETAILED DESCRIPTION:
Investigators enroll patients affected by solid tumors which present itch refractory to standard treatment ("refractory group") and patients who did not receive any treatment for pruritus ("naïve group"). The intensity of itch will be evaluated with Visual Analogue Scale (VAS) score. In the refractory group Aprepitant (125 mg on day 1; 80 mg on day 3; 80 mg on day 5) will be administered after at least 1 week of standard systemic treatment. In the naïve group, Aprepitant will be administered after the first onset of severe pruritus. The primary end point is to evaluate the effect of aprepitant in managing pruritus both in naive and refractory group.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of solid tumor
* treatment with anti-EGFR antibodies or TKIs
* first onset of severe pruritus during treatment (≥7 on Visual Analogue Scale (VAS) score)

Exclusion Criteria:

* oral treatment with antimycotics during 4 weeks preceding enrolment
* topical treatment during the previous 2 weeks
* concomitant,chronic renal or hepatic insufficiency , skin infection or dermatitis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Severity of ITCH | once before aprepitant administration; 7 days after the first dose of aprepitant, and once a week until the end of biological therapy
  Patients is asked to grade the intensity of their itch on the VAS, with the strongest possible itch marked at the right end of the line (10) and no itch marked at the left end (0). The VAS score is registered in a diary supplied 7 days before starting the study and every week throughout the study period.
  Pruritus intensity is evaluated by VAS score once before Aprepitant administration, once 7 days after the first dose of Aprepitant and once a week until the end of biological therapy or the pruritus recurrence. Response (evaluated one week after the first Aprepitant dose) is defined as > 50% reduction of pruritus intensity compared to the baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Santini, MD, PhD, Principal Investigator — Campus Bio-Medico of Rome University
Locations (1):
- Campus Bio-Medico of Rome University, Roma, Italy

REFERENCES:
- [Derived] Santini D, Vincenzi B, Guida FM, Imperatori M, Schiavon G, Venditti O, Frezza AM, Berti P, Tonini G. Aprepitant for management of severe pruritus related to biological cancer treatments: a pilot study. Lancet Oncol. 2012 Oct;13(10):1020-4. doi: 10.1016/S1470-2045(12)70373-X. Epub 2012 Sep 18. PMID 22995650